CLINICAL TRIAL: NCT02953236
Title: THE INMEDIATE EFFECTS OF RICHELLI'S PAINRELIEVER ON UPPER TRAPEZIUS MYOFASCIAL TRIGGER POINT IN PATIENTS SUFFERING FROM NECK PAIN: A RANDOMIZED CONTROLLED TRIAL
Brief Title: INSTRUMENTED-MANUAL PHYSIOTHERAPY VERSUS NONINSTRUMENTED
Acronym: ECA_TMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Principal Research PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103-2015-H
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Instrumented massage (Experimental)
  Interventions: Procedure: Instrumented massage
- Manual massage (Active Comparator)
  Interventions: Procedure: Manual massage

INTERVENTIONS:
Procedure: Instrumented massage — The first group will receive a 20 min session of instrumented massage on back and neck areas. Subjects will be in prone position and physical therapist will applied instrumental massage in a protocolised way from low back until neck muscles, both in left and right side of the body.
  Arms: Instrumented massage
Procedure: Manual massage — The second group will receive a 20 min session of manual massage on back and neck areas. Subjects will be in prone position and physical therapist will applied manual massage in a protocolised way from low back until neck muscles, both in left and right side of the body.
  Arms: Manual massage

SUMMARY:
This study aimed to verify the mechanical and clinical effects of instrumented massage on myofascial trigger points of trapezius muscle in adult subjects.

DETAILED DESCRIPTION:
Background: There are several therapies currently used to treat myofascial trigger points, including conservative and invasive techniques. It has been shown that conservative techniques including therapeutic massage, stretching, transcutaneal electrical nerve stimulation, spray and stretch, cold laser treatment, and ultrasound are the most applied treatments for myofascial pain syndrome, but no single strategy has proved to be universally successful. Instrumented massage has shown clinical effectiveness on shoulder pain, low back pain, and only one study (case report) on myofascial trigger points. This study aimed to verify the mechanical and clinical effects of instrumented massage on myofascial trigger points of trapezius muscle in adult subjects.

Methods/Design: The study includes 31 volunteers with myofascial trigger points on right trapezius muscle. Clinical and patient data were obtained from questionnaires, VAS, algometry, sono-myoelastography and myotonometry. Also, physiotherapist grip strength was measured. Subjects were randomly allocated into one of two groups: Instrumented massage or Manual massage. The intervention consisted in a single 20 minutes session of massage on the back and neck by the same therapist, depending of the group, massage was applied manually or instrumented.

ELIGIBILITY:
Inclusion Criteria:

* • To be of legal age.

  * To understand correctly Spanish.
  * To show their approval by signing the informed consent.
  * Suffering from mechanical neck pain

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
• Pain as measured by VAS | 10 minutes
  The Visual Analogue Scale (VAS) was designed to allow a subjective assessment of pain. A VAS is usually a horizontal line of 10 cm. with perpendicular lines at the ends, which are defined as the extreme limits of the painful experience. Previous studies have shown that the VAS has adequate psychometric properties, including test-retest reliability (r = 0.78) and convergent validity with other measures of pain such as the McGill Pain Questionnaire (r = 0.49 to 0.65) (Sriwatanakul K ., 1983).
• Stiffness of the right upper trapezius myofascial trigger point measured by MyoptronPRO. | 10 minutes
  Stiffness characteristics will be measured using a handheld MyotonPRO device (MyotonPRO, Myoton Ltd, Estonia). MyotonPRO has shown high levels of reliability in a session or between sessions both by the same operator (intra-rater) and between different operators (inter-rater), both in young subjects and elderly (Aird et al., 2012) (Mullix et al., 2012). Stiffness (N/m) will be calculated by software of MyotonPRO (Vain, 1994, 1995). Stiffness is the ability of tissue to restore it shape after removing of external force acting on the muscle.
• Stiffness (Hz) of the right upper trapezius myofascial trigger point measured by sono-myoelastography. | 10 minutes
  Sono-myoelastography uses an external vibration source with a frequency less than 1000 Hz in conjunction with Doppler techniques to identify localized regions of increased tissue stiffness (Muro-Culebras, 2013). In this study vibrations will be produced in the right upper trapezius muscle using an external massage vibrator (Model NC70209, North Coast Medical, Gilroy, CA, USA) modified with a flat and elongated applicator (with an application area of 1 x 4 cm). This vibration source will be placed approximately 2-3 cm away from each of the points marked as ''positive'' in the clinical examination and induce vibrations of about 92 Hz. By use of the power Doppler technique, the sono-myoelastography images will be collected while applying vibrations.

SECONDARY OUTCOMES:
pain threshold pressure PPT | 10 minutes
• Grip strength as measured by a Dynamometer | 10 minutes
  This instrument will be used to measure grip strength of both physiotherapist upper limbs. The dynamometer has proven to be the safest [ICC = 0.98] and most valid [ICC = 0.99] method to measure grip strength of the hand. (Bellace JV, 2000).
•PRO Spine Functional Index SFI-Sp | 10 minutes
  For this study we will use the Spanish version (SFI-Sp), since it has proven to be a valid and reliable measure of the spinal region result. This regional tool reflects the status and any change in the kinetic chain of the spine. This questionnaire has demonstrated high internal consistency (α = 0.85) and reliability (r = 0.96) (AI Cuesta-Vargas, 2014).
•PRO Neck Disability Index-Sp | 10 minutes
  Neck Disability Index is the most widely used neck pain scale in the largest number of populations and has been validated most often against multiple measurements of function, pain, and clinical signs and symptoms. (Cleland et al., 2006). For this study we will use the Spanish version (NDI-Sp), since it has proven to be reliable (r = 0.98), valid, and sensitive to change. (Andrade et al., 2010).
• Blood flow of the right upper trapezius myofascial trigger point measured by sono-myoelastography. | 10 minutes
  Circulation will be studied using the Doppler technique, since it has been shown for other studies (Sikdar et al., 2009). The resistive index (RI) is determined in the ascending branch of the transverse cervical artery and in other arteries or arterioles that will be in the vicinity of points marked as ''positive'' in the clinical examination. The waveform of blood flow, based on Doppler flow, will be scored on a scale of 0-2 (Sikdar et al. 2009).

OTHER OUTCOMES:
• Tone of the right upper trapezius myofascial trigger point measured by MyoptronPRO | 10 minutes
  Muscle tone characteristics will be measured using a handheld MyotonPRO device (MyotonPRO, Myoton Ltd, Estonia). Muscle tone will be calculated by software of MyotonPRO (Vain, 1994, 1995). Muscle tone (Hz) is the frequency of damped mechanical oscillation of muscle tissue, is an index of the tension in the muscle
• Elasticity of the right upper trapezius myofascial trigger point measured by MyoptronPRO | 10 minutes
  Muscle elasticity characteristics will be measured using a handheld MyotonPRO device (MyotonPRO, Myoton Ltd, Estonia). Elasticity (logarithmic decrement of oscillations amplitude damping) will be calculated by software of MyotonPRO (Vain, 1994, 1995). Elasticity is the ability of muscle to restore its initial shape after contraction. A lower level of decrement reveals a better muscle elasticity and ability of contraction.
• Morphology of the right upper trapezius myofascial trigger point measured by sono-myoelastography. | 10 minutes
  It will be obtained from a sonographic examination using the B-mode of a clinical ultrasound scanner with a linear transducer (Esaote Mylabs25, Milan, Italy) set to a frequency of 12 MHz and depth of 4 cm, since some studies have described the possibility of using sonography in the diagnosis of myofascial trigger points. (Sikdar et al., 2009). Finally, the operator will use the ''ellipse'' tool of the ultrasound to delineate and calculate the size of the largest hypoechoic area found.

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Cuesta-Vargas, Málaga, Malaga, Spain

IPD SHARING:
Plan to Share IPD: Yes